CLINICAL TRIAL: NCT00851643
Title: A Randomized, Double-Blind, Multicenter, Biphasic, Controlled With GARDASIL™ Dose-Escalation Study of Octavalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine Adjuvanted With Amorphous Aluminum Hydroxyphosphate Sulfate (AAHS) and ISCOMATRIX™ (IMX)
Brief Title: Broad Spectrum HPV Vaccine Dose Escalation Study (V502-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V502-002; 2009_552
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Human Papilloma Virus; Cervical Cancer; Vulvar Cancer; Vaginal Cancer; Genital Warts
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- qHPV (GARDASIL™) - Phase A Control (Active Comparator): Quadrivalent Human Papillomavirus (qHPV) (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™). This is the control for the Octavalent HPV with 15 mcg ISCOMATRIX™ (IMX) / Aluminum Hydroxyphosphate Sulfate (AAHS) and Octavalent HPV with 30 mcg IMX / AAHS during Phase A.
  Interventions: Biological: Comparator: Quadrivalent HPV Vaccine (qHPV), (GARDASIL™)
- Octavalent HPV with 15 mcg IMX / AAHS (Experimental): Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 Virus-Like Particle (VLP) Vaccine Adjuvanted With 281 mcg AAHS and 15 mcg IMX.
  Interventions: Biological: Octavalent HPV with 15 mcg IMX / AAHS
- Octavalent HPV with 30 mcg IMX / AAHS (Experimental): Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 VLP Vaccine Adjuvanted With 281 mcg AAHS and 30 mcg IMX.
  Interventions: Biological: Octavalent HPV with 30 mcg IMX / AAHS
- qHPV (GARDASIL™) - Phase B Control (Active Comparator): Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™). This is the control for the Octavalent HPV with 60 mcg IMX / AAHS and Octavalent HPV with 120 mcg IMX / AAHS during Phase B.
  Interventions: Biological: Comparator: Quadrivalent HPV Vaccine (qHPV), (GARDASIL™)
- Octavalent HPV with 60 mcg IMX / AAHS (Experimental): Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 VLP Vaccine Adjuvanted With 281 mcg AAHS and 60 mcg IMX.
  Interventions: Biological: Octavalent HPV with 60 mcg IMX / AAHS
- Octavalent HPV with 120 mcg IMX / AAHS (Experimental): Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 VLP Vaccine Adjuvanted With 281 mcg AAHS and 120 mcg IMX.
  Interventions: Biological: Octavalent HPV with 120 mcg IMX / AAHS

INTERVENTIONS:
Biological: Octavalent HPV with 15 mcg IMX / AAHS — 0.5-mL intramuscular injection administered at Day 1, Month 2 and Month 6
  Other Names: V502
  Arms: Octavalent HPV with 15 mcg IMX / AAHS
Biological: Octavalent HPV with 30 mcg IMX / AAHS — 0.5-mL intramuscular injection administered at Day 1, Month 2 and Month 6
  Other Names: V502
  Arms: Octavalent HPV with 30 mcg IMX / AAHS
Biological: Octavalent HPV with 60 mcg IMX / AAHS — 0.5-mL intramuscular injection administered at Day 1, Month 2 and Month 6
  Other Names: V502
  Arms: Octavalent HPV with 60 mcg IMX / AAHS
Biological: Octavalent HPV with 120 mcg IMX / AAHS — 0.5-mL intramuscular injection administered at Day 1, Month 2 and Month 6
  Other Names: V502
  Arms: Octavalent HPV with 120 mcg IMX / AAHS
Biological: Comparator: Quadrivalent HPV Vaccine (qHPV), (GARDASIL™) — 0.5-mL intramuscular injection administered at Day 1, Month 2 and Month 6
  Other Names: V502-002
  Arms: qHPV (GARDASIL™) - Phase A Control; qHPV (GARDASIL™) - Phase B Control

SUMMARY:
This study will examine the safety and tolerability of octavalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) vaccine formulated with amorphous aluminum hydroxysulfate (AAHS) and ISCOMATRIX™ (IMX). Reviews of safety and tolerability will be used to select the dose(s) of IMX for further studies of the octavalent HPV L1 VLP vaccine.

DETAILED DESCRIPTION:
The study was performed in 2 staggered phases, Phase A and Phase B. In Phase A, participants were randomized to qHPV, Octavalent HPV with 15 mcg IMX/AAHS, or Octavalent HPV with 30 mcg IMX/AAHS. After the safety for Phase A was reviewed, Phase B was initiated. In Phase B, participants were randomized to qHPV, Octavalent HPV with 60 mcg IMX/AAHS or Octavalent HPV with 120 mcg IMX/AAHS.

ELIGIBILITY:
Inclusion Criteria:

* Participant is in good physical health
* Participant has had a lifetime history of 0 to 4 sexual partners
* Females between 18-to-24 years

Exclusion Criteria:

* Participant has a history of abnormal Pap test
* Participant has a history of positive test for HPV
* Participant has a history of recent or ongoing alcohol or drug abuse
* Participant is immunocompromised or has an autoimmune condition
* Participant has received immunosuppressive therapy within a year of screening
* Participant has previously received an HPV vaccine
* Participant is pregnant
* Participant has a history of external genital/vaginal warts
* Participant is currently enrolled in a clinical trial
* Participant has a history of a severe allergic reaction that required medical attention

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 158 participants were enrolled. Of the enrolled 158 participants, 8 were screening failures. 150 participants were randomized to the base study (up to 12 months), conducted in 2 phases, Phase A and Phase B. Some participants continued in a voluntary, long-term extension of the study (up to 36 months).
Pre-assignment Details: In Phase A, participants were randomized to quadrivalent Human Papillomavirus (qHPV), Octavalent HPV with 15 mcg ISCOMATRIX™ (IMX) / Aluminum Hydroxyphosphate Sulfate (AAHS), or Octavalent HPV with 30 mcg IMX/AAHS. In Phase B, participants were randomized to qHPV, Octavalent HPV with 60 mcg IMX/AAHS or Octavalent HPV with 120 mcg IMX/AAHS.
Groups:
- qHPV (GARDASIL™) - Phase A Control: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™)- controls from Phase A. A 0.5-mL intramuscular injection was administered at Day 1, Month 2 and Month 6.
- Octavalent HPV With 15 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 Virus-Like Particle (VLP) Vaccine Adjuvanted With 281 mcg Amorphous Aluminum Hydroxyphosphate Sulfate (AAHS) and 15 mcg ISCOMATRIX™ (IMX). A 0.5-mL intramuscular injection was administered at Day 1, Month 2 and Month 6.
- Octavalent HPV With 30 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 VLP Vaccine Adjuvanted With 281 mcg AAHS and 30 mcg IMX. A 0.5-mL intramuscular injection was administered at Day 1, Month 2 and Month 6.
- qHPV (GARDASIL™) - Phase B Control: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™)- controls from Phase B. A 0.5-mL intramuscular injection was administered at Day 1, Month 2 and Month 6.
- Octavalent HPV With 60 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 VLP Vaccine Adjuvanted With 281 mcg AAHS and 60 mcg IMX. A 0.5-mL intramuscular injection was administered at Day 1, Month 2 and Month 6.
- Octavalent HPV With 120 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 VLP Vaccine Adjuvanted With 281 mcg AAHS and 120 mcg IMX. A 0.5-mL intramuscular injection was administered at Day 1, Month 2 and Month 6.
Period: Base Study (Up to 12 Months)
Arm/Group | qHPV (GARDASIL™) - Phase A Control | Octavalent HPV With 15 mcg IMX / AAHS | Octavalent HPV With 30 mcg IMX / AAHS | qHPV (GARDASIL™) - Phase B Control | Octavalent HPV With 60 mcg IMX / AAHS | Octavalent HPV With 120 mcg IMX / AAHS
Started | 15 | 30 | 30 | 15 | 30 | 30
Completed | 14 | 30 | 30 | 15 | 30 | 29
Not Completed | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1
Period: Extension Study (Up to 36 Months)
Arm/Group | qHPV (GARDASIL™) - Phase A Control | Octavalent HPV With 15 mcg IMX / AAHS | Octavalent HPV With 30 mcg IMX / AAHS | qHPV (GARDASIL™) - Phase B Control | Octavalent HPV With 60 mcg IMX / AAHS | Octavalent HPV With 120 mcg IMX / AAHS
Started | 10 | 19 | 19 | 7 | 21 | 15
Completed | 6 | 15 | 14 | 5 | 19 | 14
Not Completed | 4 | 4 | 5 | 2 | 2 | 1
Not completed — Lost to Follow-up | 4 | 2 | 4 | 1 | 2 | 0
Not completed — Moved | 0 | 2 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Octavalent HPV With 15 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 Virus-Like Particle (VLP) Vaccine Adjuvanted With 281 mcg Amorphous Aluminum Hydroxyphosphate Sulfate(AAHS) and 15 mcg ISCOMATRIX™ (IMX). A 0.5-mL intramuscular injection was administered at Day 1, Month 2 and Month 6.
- Total: Total of all reporting groups
Arm/Group | qHPV (GARDASIL™) - Phase A Control | Octavalent HPV With 15 mcg IMX / AAHS | Octavalent HPV With 30 mcg IMX / AAHS | qHPV (GARDASIL™) - Phase B Control | Octavalent HPV With 60 mcg IMX / AAHS | Octavalent HPV With 120 mcg IMX / AAHS | Total
Number analyzed (Participants) | 15 | 30 | 30 | 15 | 30 | 30 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.3 (1.6) | 20.8 (1.8) | 20.2 (1.5) | 19.9 (1.6) | 20.5 (1.8) | 20.8 (2.0) | 20.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 30 | 30 | 15 | 30 | 30 | 150
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 15 | 30 | 30 | 15 | 30 | 30 | 150

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) to Each of the HPV Types Contained in the Vaccine for Phase A
Description: The quadrivalent HPV (GARDASIL™) vaccine has types 6, 11, 16, 18, and the octavalent HPV has types 6, 11, 16, 18, 31, 45, 52, and 58. Serum antibody titres to the HPV type were obtained using a competitive Luminex immunoassay (cLIA) after vaccination with GARDASIL™ or the octavalent HPV vaccine. GMTs were calculated and are reported as the antibody concentration in milli-Merck Units per milliliter (mMU/mL) of neutralizing monoclonal antibody equivalent.
Time Frame: 4 weeks postdose 3 (Phase A)
Population: Per Protocol Immunogenicity (PPI) population: participants who were not protocol violators, received all 3 vaccinations within acceptable day ranges, were seronegative at Day 1 and polymerase chain reaction (PCR)-negative Day 1 through Month 7 for the relevant HPV type(s), had a valid Month 7 serology result collected in the appropriate day range.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- qHPV (GARDASIL™) - Phase A Control: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™) for Phase A
- Octavalent HPV With 15 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 Virus-Like Particle (VLP) Vaccine Adjuvanted With 281 mcg Amorphous Aluminum Hydroxyphosphate Sulfate (AAHS) and 15 mcg ISCOMATRIX™(IMX)
- Octavalent HPV With 30 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 Virus-Like Particle (VLP) Vaccine Adjuvanted With 281 mcg Amorphous Aluminum Hydroxyphosphate Sulfate (AAHS) and 30 mcg ISCOMATRIX™ (IMX)
Arm/Group | qHPV (GARDASIL™) - Phase A Control | Octavalent HPV With 15 mcg IMX / AAHS | Octavalent HPV With 30 mcg IMX / AAHS
Number analyzed (Participants) | 15 | 30 | 30
mMU/mL
  Anti-HPV 6 (N=11, N=21, N=22) | 1273.3 [704.9 to 2300.1] | 2203.0 [1658.9 to 2925.6] | 4784.7 [3741.5 to 6118.8]
  Anti-HPV 11 (N=11, N=21, N=22) | 1991.6 [1096.3 to 3618.2] | 2564.3 [1940.8 to 3388.3] | 3921.6 [2964.4 to 5188.0]
  Anti-HPV 16 (N=11, N=23, N=24) | 2381.9 [1558.5 to 3640.4] | 3961.8 [2982.6 to 5262.4] | 7484.4 [5493.9 to 10196.1]
  Anti-HPV 18 (N=11, N=24, N=24) | 568.7 [284.8 to 1135.7] | 1375.7 [966.4 to 1958.2] | 2315.3 [1453.4 to 3688.3]
  Anti-HPV 31(N=11, N=24, N=23) | 24.3 [NA to 79.1] — The lower bound of the 95% confidence interval is below the level of detectability (<8). | 2037.5 [1502.4 to 2763.0] | 4782.3 [3282.4 to 6967.5]
  Anti-HPV 45 (N=11, N=26, N=25) | 10.8 [NA to 52.7] — The lower bound of the 95% confidence interval is below the level of detectability (<4). | 1042.8 [760.8 to 1429.1] | 2116.5 [1329.7 to 3368.8]
  Anti-HPV 52 (N=9, N=23, N=25) | NA [NA to NA] — The lower and upper bounds of the 95% confidence interval are below the level of detectability (<16 to <16). | 2531.1 [1798.6 to 3561.9] | 4292.0 [2997.7 to 6145.2]
  Anti-HPV 58 (N=10, N=24, N=22) | 17.7 [NA to 86.1] — The lower bound of the 95% confidence interval is below the level of detectability (<6). | 1759.2 [1276.5 to 2424.4] | 3146.4 [2335.4 to 4428.8]

2. Primary Outcome: Geometric Mean Titers (GMTs) to Each of the HPV Types Contained in the Vaccine for Phase B
Description: The quadrivalent HPV (GARDASIL™) vaccine has types 6, 11, 16, 18, and the octavalent HPV has types 6, 11, 16, 18, 31, 45, 52, and 58. Serum antibody titres to the HPV type were obtained using cLIA after vaccination with GARDASIL™ or the octavalent HPV vaccine. GMTs were calculated and are reported as the antibody concentration in milli-Merck Units per milliliter (mMU/mL) of neutralizing monoclonal antibody equivalent.
Time Frame: 4 weeks postdose 3 (Phase B)
Population: PPI population: All participants who were not protocol violators, received all 3 vaccinations within acceptable day ranges, were seronegative at Day 1 and PCR-negative Day 1 through Month 7
  for the relevant HPV type(s), and had a valid Month 7 serology result collected in the appropriate day range.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- qHPV (GARDASIL™) - Phase B Control: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™) for Phase B
- Octavalent HPV With 60 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 Virus-Like Particle (VLP) Vaccine Adjuvanted With 281 mcg Amorphous Aluminum Hydroxyphosphate Sulfate (AAHS) and 60 mcg ISCOMATRIX™(IMX)
- Octavalent HPV With 120 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 Virus-Like Particle (VLP) Vaccine Adjuvanted With 281 mcg Amorphous Aluminum Hydroxyphosphate Sulfate (AAHS) and 120 mcg ISCOMATRIX™ (IMX)
Arm/Group | qHPV (GARDASIL™) - Phase B Control | Octavalent HPV With 60 mcg IMX / AAHS | Octavalent HPV With 120 mcg IMX / AAHS
Number analyzed (Participants) | 15 | 30 | 30
mMU/mL
  Anti-HPV Type 6 (N=10, N=19, N=23) | 2350.9 [1581.6 to 3494.2] | 6006.0 [3991.6 to 9037.0] | 4484.8 [2791.7 to 7204.7]
  Anti-HPV Type 11 (N=10, N=19, N=23) | 3762.2 [2422.0 to 5844.1] | 6514.2 [4520.8 to 9386.8] | 6609.3 [5028.2 to 8687.5]
  Anti-HPV Type 16 (N=7, N=19, N=20) | 2783.6 [973.2 to 7961.8] | 12947.5 [8856.5 to 18928.3] | 10105.9 [6570.9 to 15542.6]
  Anti-HPV Type 18 (N=10, N=19, N=25) | 948.2 [403.7 to 2227.1] | 5090.0 [3467.5 to 7471.7] | 4070.9 [3135.2 to 5285.9]
  Anti-HPV Type 31 (N=11, N=22, N=24) | 36.9 [15.5 to 88.2] | 7779.0 [4876.7 to 12408.5] | 5487.3 [3683.0 to 8175.6]
  Anti-HPV Type 45 (N=11, N=20, N=24) | 4.7 [NA to 10.9] — The lower bound of the 95% confidence interval is below the level of detectability (<4). | 3974.8 [2680.5 to 5894.0] | 4696.4 [3499.6 to 6302.5]
  Anti-HPV Type 52 (N=10, N=20, N=23) | NA [NA to NA] — The GMT is <16, and the lower and upper bounds of the 95% confidence interval are below the level of detectability (<16 to <16). | 5714.9 [3962.4 to 8242.6] | 6624.6 [4919.9 to 8919.9]
  Anti-HPV Type 58 (N=9, N=21, N=24) | 9.6 [NA to 28.1] — The lower bound of the 95% confidence interval is below the level of detectability (<6). | 4961.8 [3170.1 to 7766.1] | 5191.2 [4036.3 to 6676.5]

3. Primary Outcome: Number of Participants Who Seroconverted to Each of the HPV Types Contained in the Vaccine During Phase A
Description: A vaccinated participant was considered seropositive for a given HPV type if her serum antibody titer by cLIA for the HPV type was greater than the serostatus cutoff. The serostatus cutoffs for HPV Types 6, 11, 16, 18, 31, 45, 52, and 58 were 20, 20, 20, 20, 16, 16, 20, and 16 mMU/mL, respectively.
Time Frame: 4 weeks postdose 3 (Phase A)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | qHPV (GARDASIL™) - Phase A Control | Octavalent HPV With 15 mcg IMX / AAHS | Octavalent HPV With 30 mcg IMX / AAHS
Number analyzed (Participants) | 15 | 30 | 30
Participants
  Anti-HPV 6 (N=11, N=21, N=22) | 11 | 21 | 22
  Anti-HPV 11 (N=11, N=21, N=22) | 11 | 21 | 22
  Anti-HPV 16 (N=11, N=23, N=24) | 11 | 23 | 24
  Anti-HPV 18 (N=11, N=24, N=24) | 11 | 24 | 24
  Anti-HPV 31 (N=11, N=24, N=23) | 6 | 24 | 23
  Anti-HPV 45 (N=11, N=26, N=25) | 4 | 26 | 25
  Anti-HPV 52 (N=9, N=23, N=25) | 0 | 23 | 25
  Anti-HPV 58 (N=10, N=24, N=22) | 3 | 24 | 22

4. Primary Outcome: Number of Participants Who Seroconverted to Each of the HPV Types Contained in the Vaccine During Phase B
Description: as for outcome 3
Time Frame: 4 weeks postdose 3 (Phase B)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | qHPV (GARDASIL™) - Phase B Control | Octavalent HPV With 60 mcg IMX / AAHS | Octavalent HPV With 120 mcg IMX / AAHS
Number analyzed (Participants) | 15 | 30 | 30
Participants
  Anti-HPV 6 (N=10, N=19, N=23) | 10 | 19 | 23
  Anti-HPV 11 (N=10, N=19, N=23) | 10 | 19 | 23
  Anti-HPV 16 (N=7, N=19, N=20) | 7 | 19 | 20
  Anti-HPV 18 (N=10, N=19, N=25) | 10 | 19 | 25
  Anti-HPV 31 (N=11, N=22, N=24) | 9 | 22 | 24
  Anti-HPV 45 (N=11, N=20, N=24) | 2 | 20 | 24
  Anti-HPV 52 (N=10, N=20, N=23) | 0 | 20 | 23
  Anti-HPV 58 (N=9, N=21, N=24) | 2 | 21 | 24

ADVERSE EVENTS:
Time Frame: All injection site adverse events (AEs) for 5 days following vaccination, all non-injection site AEs for 14 calendar days following vaccination, and all laboratory AEs that occurred at any time during the study are included.
Groups:
- qHPV (GARDASIL™) - Phase A and Phase B Controls: Quadrivalent Human Papillomavirus (qHPV) (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™) combined from Phase A and Phase B.
- Octavalent HPV With 15 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 VLP vaccine adjuvanted with 281 mcg AAHS and 15 mcg IMX.
- Octavalent With 120 mcg IMX / AAHS: Octavalent Human Papillomavirus (HPV) (Types 6, 11, 16, 18, 31, 45, 52, and 58) L1 VLP vaccine adjuvanted with 281 mcg AAHS and 120 mcg IMX.
Arm/Group | qHPV (GARDASIL™) - Phase A and Phase B Controls | Octavalent HPV With 15 mcg IMX / AAHS | Octavalent HPV With 30 mcg IMX / AAHS | Octavalent HPV With 60 mcg IMX / AAHS | Octavalent With 120 mcg IMX / AAHS
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30 | 30/30 | 30/30 | 30/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV (GARDASIL™) - Phase A and Phase B Controls (N=30) | Octavalent HPV With 15 mcg IMX / AAHS (N=30) | Octavalent HPV With 30 mcg IMX / AAHS (N=30) | Octavalent HPV With 60 mcg IMX / AAHS (N=30) | Octavalent With 120 mcg IMX / AAHS (N=30)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 2 (2) | 2 (4) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 5 (6) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 2 (2) | 6 (11) | 6 (6) | 9 (10)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Axillary pain (General disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (5) | 2 (3)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 4 (4) | 1 (1) | 3 (4) | 1 (1)
Injection site erythema (General disorders) | 12 (21) | 15 (18) | 16 (27) | 21 (36) | 20 (38)
Injection site haematoma (General disorders) | 1 (1) | 2 (3) | 7 (7) | 3 (3) | 4 (5)
Injection site induration (General disorders) | 0 (0) | 4 (6) | 5 (8) | 5 (10) | 5 (6)
Injection site mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 4 (5)
Injection site pain (General disorders) | 27 (62) | 29 (94) | 30 (101) | 30 (95) | 30 (89)
Injection site pruritus (General disorders) | 3 (5) | 4 (6) | 1 (1) | 5 (7) | 5 (7)
Injection site swelling (General disorders) | 7 (14) | 15 (22) | 22 (37) | 24 (48) | 22 (43)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 1 (1) | 5 (5) | 12 (15)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 0 (0) | 3 (4) | 3 (3) | 3 (3)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 4 (4) | 5 (5)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 4 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 4 (4) | 2 (2) | 3 (5)
Headache (Nervous system disorders) | 12 (22) | 10 (16) | 16 (29) | 15 (30) | 19 (46)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (7) | 1 (1) | 3 (3) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As this study is part of a multicenter trial, the SPONSOR does not recommend separate publication of individual study site results due to scientific concerns. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.